CLINICAL TRIAL: NCT05048992
Title: Effects of ElDOA and Post-Facilitation Stretching Technique on Pain and Disability in Patients With Text Neck Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCE/Lhr/0116 Maryam
Record Dates: First submitted 2021-09-13; First posted 2021-09-17 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Neck Pain
Keywords: Text Neck Syndrome
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ELDOA method (Active Comparator): Twenty (20) patients will be treated with ELDOA method
  Interventions: Other: ELDOA method
- Post-facilitation stretching (Active Comparator): Twenty (20) patients will be treated with Post-facilitation stretching technique.
  Interventions: Other: Post-facilitation stretching

INTERVENTIONS:
Other: ELDOA method — group A will receive
  Arms: ELDOA method
Other: Post-facilitation stretching — Group B will receive
  Arms: Post-facilitation stretching

SUMMARY:
In this modern era, Text Neck is a new term used to describe neck pain and associated damage caused by continuous flexed posture due to excessive use of smartphones for a long time. The term text neck was first introduced by Dr. Dean L. Fishman, who is US based chiropractor. Text neck can also be described as overuse syndrome caused by repetitive stress on neck due to prolonged flexion. There is coordinated work between cervical spine and surrounding structure such as muscles, ligament, nerves and bones. In addition, any nerve compression at cervical spine leads to radiating pain in neck, shoulder and arm. Previous literature reported use of cell phone is very common in population of 18 to 44 years of age. Seventy nine percent (79%) population have smartphone with them all the time. Technology has become essential part of modern lifestyle. Sustained flexed posture forces the head to exert weight on neck of varying degrees. Weight of neutral head is 10 to 12 pounds and increases 6 times 1 inch forward movement of head. Children are at higher risk because of their large head size. This study will be a Randomized clinical trial with objective to reduce neck pain and disability in patients with text neck syndrome. Two groups will be designed, in one group ElDOA (n=20) and in other group post facilitation technique (n=20) will be applied. Patients will be recruited into two groups by consecutive sampling by non-replacement lottery method with equal no. of chits. Patients will be assessed by Numeric pain rating scale (NPRS), Neck disability index (NDI), smartphone addiction scale before and after treatment. Both groups will receive heating pad as common treatment first after that group A will be treated with ELDOA and group B will be treated with Post-facilitation. Session of 6 weeks with 3 days per week will be conducted. After that post treatment assessment will be done.

ELIGIBILITY:
Inclusion Criteria:

* • Neck pain without unilateral UE symptoms

  * Age 18-35 years
  * Subjects using Phone since past 1 year
  * Neck disability index (NDI) score >10 points
  * Participants able to understand and fill the questionnaire in English

Exclusion Criteria:

* • Subjects having any congenital cervical condition

  * Subjects having traumatic cervical condition such as whiplash injury within the past 6 weeks
  * History of spinal tumors, spinal infection, cervical spine fracture, or previous neck surgery
  * Subjects with cervical radiculopathy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-30 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 6 weeks
  will be used for pain measurement. It is a uni-dimensional 11 point scale (0-10) with measure of pain intensity.
Neck disability index (NDI) | 6 weeks
  ) will be used to assess neck disability. It consists of 10 sections and each section carries 5 marks. 0 indicate no activity limitation and 5 indicates complete activity limitation.
Smartphone addiction scale (SAS) | 6 weeks
  will be used to assess smartphone addiction. It is self-reporting scale consist of 6 factors and 33 items. Score ranges from 33 to 198 and higher the score greater the degree of addiction.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Salman Bashir, PhD, Principal Investigator — Riphah International University
Locations (1):
- Safi Hospital Faisalabad, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee JI, Song HS. The correlation analysis between hours of smartphone use and neck pain in the Gachon university students. Journal of Acupuncture Research. 2014;31(2):99-109.
- [Background] Neupane S, Ali U, Mathew A. Text neck syndrome-systematic review. Imperial Journal of Interdisciplinary Research. 2017;3(7):141-8
- [Background] Vate-U-Lan P. Text neck epidemic: a growing problem for smart phone users in Thailand. International Journal of the Computer, the Internet and Management. 2015;23(3):551-6.